CLINICAL TRIAL: NCT03776864
Title: A Phase II Trial of Umbralisib and Pembrolizumab in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Umbralisib and Pembrolizumab in Treating Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company providing drug terminated their oncology program
Sponsor: University of Washington (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Ryan Lynch, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1003718; NCI-2018-02836 (Other: NCI / CTRP); 10075 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab; Immunoglobulin G; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, umbralisib) (Experimental): Patients receive pembrolizumab IV on day 1. Treatment repeats every 21 for up to 16 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive umbralisib PO daily on days 1-21 days. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Umbralisib

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Immunoglobulin G4; Anti-(Human Programmed Cell Death 1); Lambrolizumab; MK-3475; SCH 900475
Drug: Umbralisib — Given PO
  Other Names: TGR-1202; RP5264

SUMMARY:
This phase II trial studies how well umbralisib and pembrolizumab work in treating patients with classical Hodgkin lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Umbralisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Giving umbralisib and pembrolizumab may work better in treating classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive pembrolizumab IV on day 1. Treatment repeats every 21 for up to 16 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive umbralisib orally (PO) daily on days 1-21 days. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days, then up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CHL that has received at least 1 prior lines of therapy
* Measurable fludeoxyglucose F-18 (FDG)-avid disease defined by standard criteria (Lugano 2014) and a minimum of 1.0 cm in diameter
* Prior treatment with anti-PD1 or anti-PDL1 therapy is allowed.

  * Patients who are currently on anti-PD1 or anti-PDL1 therapy who have failed to achieve a CR after at least 18 weeks of treatment may enroll on study. For these patients, anti-PD1 or anti-PDL1 therapy may be delayed for screening and to align pembrolizumab dosing with the expected cycle 1 day 1. Patients with progressive disease after prior anti-PD1 or anti-PDL1 therapy do not have to be treated for 18 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Ability to swallow and retain oral medication
* Willingness and ability to comply with study and follow-up procedures, and give written informed consent
* Female subjects of childbearing potential must be surgically sterile, be post-menopausal (for at least 1 year prior to screening visit), or must have a negative pregnancy test within 3 days prior to cycle 1 day 1 and agree to use medically acceptable contraception throughout the study period and for 4 months after the last dose of either study drug. Men of reproductive potential may not participate unless they agree to use medically acceptable contraception throughout the study period and for 4 months after the last dose of either study drug
* Patients must be expected to receive at least 2 cycles of therapy
* Patients should have a life expectancy if untreated of >= 90 days in the opinion of the investigator
* Patients must have a FDG-positron emission tomography (PET)-computed tomography (CT) of chest, abdomen, and pelvis within 42 days of enrollment
* Absolute neutrophil count (ANC) > 750
* Platelet count > 40,000
* Total bilirubin =< 1.5 times the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (if known liver involvement then =< 5 x ULN is allowed)
* Calculated creatinine clearance > 30 mL/min (as calculated by the Cockcroft-Gault formula)

Exclusion Criteria:

* Patients receiving cancer therapy (i.e., chemotherapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization, prednisone > 10 mg or equivalent) or any investigational drug within 21 days of cycle 1 day 1. Patients receiving radiation therapy within 14 days from cycle 1 day 1. Anti-PD1 or anti-PDL1 therapy in patients with less than a CR after 18 weeks of such therapy is permitted to continue on schedule
* Discontinuation from prior anti-PD1 or anti-PDL1 therapy due to immune-related adverse event or any other treatment-related adverse event
* Autologous transplantation within 100 days
* Prior allogeneic transplant within 12 months of initiation on study
* Active graft versus host disease (GVHD) within 90 days prior to cycle 1 day 1
* Evidence of active central nervous system lymphoma
* Pregnant or nursing women
* Evidence of chronic active hepatitis B or chronic active hepatitis C infection (hepatitis C virus [HCV]), active cytomegalovirus (CMV), or known history of human immunodeficiency virus (HIV). If hepatitis B core (HBc) antibody, HCV antibody or CMV immunoglobulin (Ig)M is positive, the patient should be correspondingly evaluated for the presence of HBV, HCV or CMV by deoxyribonucleic acid (DNA) (polymerase chain reaction [PCR]) to determine presence or absence of active infection. If HBc antibody is positive, the subject must be evaluated for the presence of hepatitis B virus (HBV) DNA by polymerase chain reaction (PCR). If HCV antibody is positive, the subject must be evaluated for the presence of HCV ribonucleic acid (RNA) by PCR. Subjects with positive HBc antibody and negative HBV DNA by PCR are eligible. Subjects with positive HCV antibody and negative HCV RNA by PCR are eligible. Subjects who are cytomegalovirus (CMV) IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible
* Prior exposure to idelalisib (CAL-101), duvelisib (IPI-145), or any drug that specifically inhibits phosphoinositide-3-kinase (PI3K)
* Evidence of ongoing active systemic bacterial, fungal or viral infection
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic, or history of documented congestive heart failure (New York [NY] Heart Association functional classification III-IV)
  * Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of randomization
  * Concomitant use of medication known to cause QT prolongation or torsades de pointes. Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac/vascular stenting within 3 months of randomization
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater, unless approved by the protocol principal investigator
* Patients with an active autoimmune disorder (with the exception of autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura [ITP] or vitiligo)
* History of non-infectious pneumonitis related to prior line of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lynch, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Umbralisib)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Umbralisib)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 46 [30 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Proportion of subjects with relapsed/ refractory classical Hodgkin Lymphoma (CHL) who achieve a complete response (CR) with a regimen of umbralisib (oral, daily) and pembrolizumab (IV, day 1 of 21-day cycles). Per Response Evaluation Criteria Lugano 2014 for target lesions and assessed by PET-CT, Complete Metabolic Response (CMR), Deaville score of 1, 2, or 3 in nodal or extranodal sites with or without residual mass.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Umbralisib)
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Overall Response Rate
Description: Proportion of subjects with relapsed/ refractory classical Hodgkin Lymphoma (CHL) who achieve an overall response (OR) with a regimen of umbralisib (oral, daily) and pembrolizumab (IV, day 1 of 21-day cycles). Per Response Evaluation Criteria Lugano 2014 for target lesions and assessed by PET-CT, Complete Metabolic Response (CMR), Deaville score of 1, 2, or 3 in nodal or extranodal sites with or without residual mass; Partial Metabolic Response, Deauville score of 4 or 5 with reduced uptake compared to baseline and residual mass(es) of any size; No Response or Stable Disease, Deauville score of 4 or 5 with no significant change in FDG uptake from baseline at interim or end of treatment.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Umbralisib)
Number analyzed (Participants) | 6
Participants | 3

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Measured via CTCAE v4.0. Incidence of adverse events is defined as the count of participants who experienced an adverse event.
Time Frame: Up to 28 days post-treatment, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Umbralisib)
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse were collected from the time of informed consent through 28 days after last dose of study drug. Adverse events were collected for 2 years.
Arm/Group | Treatment (Pembrolizumab, Umbralisib)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Umbralisib) (N=6)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Alanine aminotransferase increased (Investigations) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Lightheadedness (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1)
Frequent urination (Renal and urinary disorders) | 1 (1)
Difficulty urinating (Renal and urinary disorders) | 1 (1)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (2)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Palate lesion (General disorders) | 1 (1)
Allergies (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Bilateral axilla pain (General disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cramping in legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Bitter taste in mouth (Gastrointestinal disorders) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Perceived distal vascular insufficiency (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT03776864/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT03776864/ICF_000.pdf